CLINICAL TRIAL: NCT01088048
Title: A Phase I Study to Investigate the Safety and Clinical Activity of Idelalisib in Combination With Chemotherapeutic Agents, Immunomodulatory Agents and Anti-CD20 mAb in Subjects With Relapsed or Refractory Indolent B-cell Non-Hodgkin Lymphoma, Mantle Cell Lymphoma or Chronic Lymphocytic Leukemia
Brief Title: Study to Investigate Idelalisib in Combination With Chemotherapeutic Agents, Immunomodulatory Agents and Anti-CD20 Monoclonal Antibody (mAb) in Participants With Relapsed or Refractory Indolent B-cell Non-Hodgkin's Lymphoma, Mantle Cell Lymphoma or Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101-07
Record Dates: First submitted 2010-03-12; First posted 2010-03-17 (Estimated); Results first posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-02

CONDITIONS: Indolent Non-Hodgkin's Lymphoma; Chronic Lymphocytic Leukemia; Mantle Cell Lymphoma
Keywords: phosphatidylinositol 3-kinase; Ofatumumab; indolent non-Hodgkin lymphoma (iNHL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell | interventions — idelalisib; Rituximab; Bendamustine Hydrochloride; ofatumumab; fludarabine; fludarabine phosphate; Everolimus; Bortezomib; Chlorambucil; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Idelalisib + Rituximab (Experimental): Participants with chronic lymphocytic leukemia (CLL) and indolent non-Hodgkin lymphoma (iNHL) will receive treatments as follows:
  Cohort 1a: Idelalisib (IDELA) 100 mg orally twice daily (BID) on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 intravenously (IV) on Days 1, 8, 15 & 22, Cycles 1 & 2
  Cohort 2a: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Days 1, 8, 15, & 22, Cycles 1 & 2
  Cohort 3e: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Days 1, 8, 15, & 22, Cycles 1 & 2
  Cohort 4a: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle, starting Cycle 2 Day 1 with the 5th dose of rituximab + rituximab 375 mg/m^2 IV on Days 1, 8, 15, & 22, Cycles 1 & 2
  Interventions: Drug: Idelalisib; Drug: Rituximab
- Idelalisib + Rituximab + Bendamustine (Experimental): Participants with CLL, iNHL and mantle cell lymphoma (MCL) will receive treatments as follows:
  Cohort 3a: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Day 1 of each 28-day cycle, Cycles 1 - 6 + bendamustine 90 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
  Cohort 3b: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Day 1 of each 28-day cycle, Cycles 1 - 6 + bendamustine 70 mg/m^2 IV on Days 1 & 2 of each 28-day cycle from Cycles 1 - 6
  Cohort 5c: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Day 1 of each 28-day cycle, Cycles 1 - 6 + bendamustine 90 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
  Interventions: Drug: Idelalisib; Drug: Rituximab; Drug: Bendamustine
- Idelalisib + Bendamustine (Experimental): Participants with CLL and iNHL will receive treatments as follows:
  Cohort 1b: IDELA 100 mg orally BID on Days 1 - 28 of each 28-day cycle + bendamustine 90 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
  Cohort 2b: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + bendamustine 90 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
  Cohort 3f: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + bendamustine 90 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
  Cohort 3g: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + bendamustine 70 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
  Cohort 4b: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle starting Cycle 2, Day 3 (after the Cycle 2 bendamustine dosing) + bendamustine 90 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
  Interventions: Drug: Idelalisib; Drug: Bendamustine
- Idelalisib + Ofatumumab (Experimental): Participants with CLL will receive treatments as follows:
  Cohort 3c: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + ofatumumab 12 doses (300 mg (Day 1 or Day 2, Dose 1), followed 1 week later by 1,000 mg weekly for 7 doses (Doses 2 - 8), followed 5 weeks later by 1,000 mg every 4 weeks for 4 doses (Doses 9 - 12))
  Interventions: Drug: Idelalisib; Drug: Ofatumumab
- Idelalisib + Fludarabine (Experimental): Participants with CLL will receive treatments as follows:
  Cohort 3d: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + fludarabine 40 mg/m^2 orally on Days 1 - 5 of each 28-day cycle, Cycles 1 - 6
  Interventions: Drug: Idelalisib; Drug: Fludarabine
- Idelalisib + Everolimus (Experimental): Participants with MCL will receive treatments as follows:
  Cohort 5a: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + everolimus 10 mg orally once daily on Days 1 - 28 of each 28-day cycle
  Interventions: Drug: Idelalisib; Drug: Everolimus
- Idelalisib + Bortezomib (Experimental): Participants with MCL will receive treatments as follows:
  Cohort 5b: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + bortezomib 1.3 mg/m^2 subcutaneously on Days 1, 8 & 15 of each 28-day cycle
  Interventions: Drug: Idelalisib; Drug: Bortezomib
- Idelalisib + Chlorambucil (Experimental): Participants with CLL will receive treatments as follows:
  Cohort 6a: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + chlorambucil 10 mg/m^2 orally once daily for 7 days every 28 days, Cycles 1 - 12
  Interventions: Drug: Idelalisib; Drug: Chlorambucil
- Idelalisib + Rituximab + Chlorambucil (Experimental): Participants with CLL will receive treatments as follows:
  Cohort 6b: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Day 1 of each 28-day cycle, Cycles 1 - 6 + chlorambucil 10 mg/m^2 orally once daily for 7 days every 28 days, Cycles 1 - 12
  Interventions: Drug: Idelalisib; Drug: Rituximab; Drug: Chlorambucil
- Idelalisib + Rituximab + Lenalidomide (Experimental): Participants with CLL and iNHL will receive treatments as follows:
  Cohort 7a: IDELA 150 mg orally BID on Days 1 - 35 of Cycle 1 (35 days) & Days 1 - 28 of all subsequent 28-day cycles + rituximab 375 mg/m^2 IV on Days 1 & 8 of Cycle 1 & Day 1 of Cycles 2 - 6 + lenalidomide 5 mg orally once daily on Days 8 - 28 of Cycle 1 (35 days) & Days 1 - 21 of next five 28-day cycles
  Cohort 7b: IDELA 150 mg orally BID on Days 1 - 35 of Cycle 1 (35 days) & Days 1 - 28 of all subsequent 28-day cycles + rituximab 375 mg/m^2 IV on Days 1 & 8 of Cycle 1 & Day 1 of Cycles 2 - 6 + lenalidomide 10 mg orally once daily on Days 8 - 28 of Cycle 1 (35 days) & Days 1 - 21 of next five 28-day cycles
  Cohort 7c: IDELA 150 mg orally BID on Days 1 - 35 of Cycle 1 (35 days) & Days 1 - 28 of all subsequent 28-day cycles + rituximab 375 mg/m^2 IV on Days 1 & 8 of Cycle 1 & Day 1 of Cycles 2 - 6 + lenalidomide 20 mg orally once daily on Days 8 - 28 of Cycle 1 (35 days) & Days 1 - 21 of next five 28-day cycles
  Interventions: Drug: Idelalisib; Drug: Rituximab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Idelalisib — Idelalisib tablet administered orally
  Other Names: GS-1101; CAL-101; Zydelig®
Drug: Rituximab — Rituximab administered intravenously
  Other Names: Rituxan
  Arms: Idelalisib + Rituximab; Idelalisib + Rituximab + Bendamustine; Idelalisib + Rituximab + Chlorambucil; Idelalisib + Rituximab + Lenalidomide
Drug: Bendamustine — Bendamustine administered intravenously
  Other Names: Treanda
  Arms: Idelalisib + Bendamustine; Idelalisib + Rituximab + Bendamustine
Drug: Ofatumumab — Ofatumumab administered intravenously
  Other Names: Arzerra
  Arms: Idelalisib + Ofatumumab
Drug: Fludarabine — Fludarabine administered orally
  Other Names: Fludara
  Arms: Idelalisib + Fludarabine
Drug: Everolimus — Everolimus administered orally twice daily until disease progression
  Other Names: Afinitor; RAD-001
  Arms: Idelalisib + Everolimus
Drug: Bortezomib — Bortezomib administered as a subcutaneous injection
  Other Names: Velcade; codenamed PS-341
  Arms: Idelalisib + Bortezomib
Drug: Chlorambucil — Chlorambucil administered on Days 1-7 every 28 days to allow appropriate therapy for participants with CLL and to coordinate into a cycle period equivalent to other study treatment regimens.
  Other Names: Leukeran
  Arms: Idelalisib + Chlorambucil; Idelalisib + Rituximab + Chlorambucil
Drug: Lenalidomide — Lenalidomide administered orally
  Other Names: Revlimid
  Arms: Idelalisib + Rituximab + Lenalidomide

SUMMARY:
The primary objective of the study is to evaluate the safety of idelalisib in combination with an anti-CD20 monoclonal antibody (mAb), a chemotherapeutic agent, a mammalian target of rapamycin (mTOR) inhibitor, a protease inhibitor, an antiangiogenic agent, and/or an immunomodulatory agent in participants with relapsed or refractory indolent B-cell non-Hodgkin lymphoma (NHL), mantle cell lymphoma (MCL), or chronic lymphocytic leukemia (CLL).

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18
* Previously treated with relapsed or refractory disease (refractory defined as not responding to a standard regimen or progressing within 6 months of the last course of a standard regimen)
* Disease status requirement:

  * For CLL patients, symptomatic disease that mandates treatment as defined by the International Workshop on Chronic Lymphocytic Lymphoma (IWCLL) 2008 criteria
  * For indolent NHL and MCL patients, measurable disease by CT scan defined as at least 1 lesion that measures > 2 cm in a single dimension
* WHO performance status of ≤ 2
* For men and women of child-bearing potential, willing to use adequate contraception (ie, latex condom, cervical cap, diaphragm, abstinence, etc.) for the entire duration of the study.

  * For Cohort 7 only: Women of child bearing potential must have 2 negative pregnancy tests prior to starting lenalidomide.
* Able to provide written informed consent

Key Exclusion Criteria:

* Is not a good candidate to receive any of the drugs administered in the study for a given disease (idelalisib, bendamustine, rituximab, ofatumumab, fludarabine, everolimus, bortezomib, or chlorambucil), according to the clinical judgment of the investigator
* Patients with atypical immunophenotype with t(11:14) translocation or cyclin D1 over-expression (CLL patients only)
* Had radiotherapy, radioimmunotherapy, biological therapy, chemotherapy, or treatment with an investigational product within 4-weeks prior to the baseline disease status tests
* Had treatment with a short course of corticosteroids for symptom relief within 1-week prior to the baseline disease status tests
* Has had an allogeneic hematopoietic stem cell transplant
* Has known active central nervous system involvement of the malignancy
* Is pregnant or nursing
* Has active, serious infection requiring systemic therapy. Patients may receive prophylactic antibiotics and antiviral therapy at the discretion of the investigator
* Has absolute neutrophil count (ANC) < 1000/µL, unless it is related to underlying CLL, MCL or indolent NHL, the latter documented by > 50% infiltration of bone marrow by tumor cells
* Has platelet count < 75000/µL, unless it is related to underlying CLL, MCL, or iNHL, the latter documented by > 50% infiltration of bone marrow by tumor cells
* Has serum creatinine ≥ 2.0 mg/dL

  * For Cohort 7 only: Has creatinine clearance < 60 mL/min
* Has serum bilirubin ≥ 2 mg/dL (unless due to Gilbert's syndrome) for patients with iNHL or CLL; for patients with MCL, serum bilirubin ≥ 1.5 x upper limit of normal
* Has serum aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≥ 2 x upper limit of normal
* Has Child-Pugh Class B or C hepatic impairment
* Has a positive test for HIV antibodies
* Has active hepatitis B or C (confirmed by RNA test). Patients with serologic evidence of prior exposure are eligible.
* Prior treatment with idelalisib

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2010-03-25 (Actual); Primary Completion 2015-04-28 (Actual); Study Completion 2015-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (11):
- United States (11):
  - Clearview Cancer Institute, Huntsville, Alabama
  - UCLA, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Weill Medical College of Cornell, New York, New York
  - Willamette Valley Cancer Institute and Research Center, Springfield, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer, Houston, Texas
  - North Star Lodge Cancer Center, Yakima, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Result] Barrientos JC, Coutre SE, de Vos S, et al. Long-term follow-up of a Phase 1b trial of idelalisib in combination with chemoimmunotherapy in patients with relapsed/refractory chronic lymphocytic leukemia including patients with del17p/TP53 mutation. 51st Annual Meeting of the American Society of Clinical Oncology (ASCO). 29 May-02 June 2015; Chicago, IL, USA. [Poster 7011].
- [Result] Barrientos J, Coutre S, de Vos S, et al. Long-term follow-up of a Phase 1 study evaluating the selective PI3K-delta inhibitor idelalisib in combination with bendamustine (B), bendamustine/rituximab (BR), fludarabine (F), chlorambucil (Chl), Or chlorambucil/rituximab (ChlR) in patients with relapsed or refractory chronic lymphocytic leukemia. Society of Hematology (ASH) Annual Meeting. December 6-9, 2014; San Francisco, CA, USA. Poster 3343.
- [Result] de Vos S, Wagner-Johnston N, Coutre S, et al. Durable responses following treatment with the PI3K-delta inhibitor idelalisib in combination with rituximab, bendamustine, or both, in recurrent indolent non-Hodgkin lymphoma: Phase I/II results. Society of Hematology (ASH) Annual Meeting. December 6-9, 2014; San Francisco, CA, USA. Poster 3063.
- [Result] Barrientos J, Leonard J, Furman R, Flinn I, De Vos S, Coutre S, et al. Phase 1b study of idelalisib (GS-1101) plus chlorambucil ± rituximab in patients with relapsed and refractory chronic lymphocytic leukemia (CLL). European Hematology Association (EHA) 2013 Congress, 13-16 June 2013; Stockholm, Sweden. Abstract P100.
- [Result] Barrientos J, Sharman J, De Vos S, et al. GS-1101 (CAL-101), selective phosphatidylinositol 3-Kinase inhibitor, in combination with ofatumumab for treatment of relapsed/refractory chronic lymphocytic leukemia. European Hematology Association (EHA) 2012 Congress, 14-17 June 2012; Amsterdam, The Netherlands. Abstract 1062.
- [Result] Coutre S, Leonard J, Furman R, et al. Combinations of the selective phosphatidylinositol 3 Kinase-delta (PI3Kd) inhibitor GS-1101 (CAL-101) with rituximab and/or bendamustine are tolerable and highly active in patients with relapsed or refractory chronic lymphocytic leukemia (CLL): results from a phase 1 study. American Society of Hematology (ASH) Annual Meeting. 8-11 December 2012; Atlanta, GA, USA. Abstract 642.
- [Result] de Vos S, Schreeder M, Finn I, et al. A phase 1 study of the selective phosphatidylinositol 3 Kinase-delta (PI3Kd) inhibitor CAL-101 (GS-1101) in combination with rituximab and/or bendamustine in patients with relapsed or refractory indolent non-Hodgkin lymphoma (iNHL). American Society of Hematology (ASH) 2011 Annual Meeting, 10-13 December 2011; San Diego, CA, USA. Abstract 2699.
- [Result] Flinn I, Schreeder M, Wagner-Johnson N, et al. A phase 1 study of CAL-101, an isoform-selective inhibitor of phosphatidylinositol 3-Kinase P110δ, in combination with rituximab and/or bendamustine in patients with relapsed or refractory B-cell malignancies. American Society of Hematology (ASH) 2010 Annual Meeting, 04-07 December 2010; Orlando, FL, USA. Blood (ASH Annual Meeting Abstracts) 2010 116: Abstract 2832.
- [Result] Flinn I, Schreeder M, Coutre S, et al. A phase 1 study of CAL-101, an isoform-selective inhibitor of phosphatidylinositol 3-Kinase P110δ, in combination with anti-CD20 monoclonal antibody therapy and/or bendamustine in patients with previously treated B-cell malignancies. 47th Annual Meeting of the American Society of Clinical Oncology (ASCO). 04-08 June 2011; Chicago, IL, USA. [Poster 3064].
- [Result] Fowler N, de Vos S, Schreeder M, et al. Combinations of the phosphatidylinositol 3 Kinase delta (PI3Kd) inhibitor idelalisib (GS-1101) with rituximab and/or bendamustine are tolerable and highly active in previously treated, indolent non-Hodgkin lymphoma: results from a phase 1 study. American Society of Hematology (ASH) 2012.
- [Result] Furman R, Barrientos J, Sharman J, et al. A phase 1/2 study of the selective phosphatidylinositol 3-Kinase-delta (PI3Kd) inhibitor CAL-101 (GS-1101) with ofatumumab in patients with previously treated chronic lymphocytic leukemia (CLL). [Poster 6518] 2012 American Society of Clinical Oncology (ASCO) Annual Meeting; 01 05 June, 2012; Chicago, IL, USA. Gilead Sciences, Inc. [Poster 6518].
- [Result] Sharman J, de Vos S, Leonard J, et al. A phase 1 study of the selective phosphatidylinositol 3-Kinase-delta (PI3Kd) inhibitor CAL-101 (GS-1101) in combination with rituximab and/or bendamustine in patients with relapsed or refractory chronic lymphocytic leukemia. American Society of Hematology (ASH) 2011 Annual Meeting, 10-13 December 2011; San Diego, CA, USA. Abstract 1787.
- [Result] Wagner-Johnston ND, De Vos S, Leonard J, Sharman JP, Schreeder MT, Boccia RV, et al. Preliminary results of PI3Kδ inhibitor idelalisib (GS-1101) treatment in combination with everolimus, bortezomib, or bendamustine/rituximab in patients with previously treated mantle cell lymphoma (MCL) [Abstract 8501]. J Clin Oncol (ASCO Annual Meeting Abstracts) 2013;31 (suppl).
- [Derived] Coutre SE, Flinn IW, de Vos S, Barrientos JC, Schreeder MT, Wagner-Johnson ND, Sharman JP, Boyd TE, Fowler N, Dreiling L, Kim Y, Mitra S, Rai K, Leonard JP, Furman RR. Idelalisib in Combination With Rituximab or Bendamustine or Both in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia. Hemasphere. 2018 Apr 25;2(3):e39. doi: 10.1097/HS9.0000000000000039. eCollection 2018 Jun. PMID 31723767
- [Derived] de Vos S, Wagner-Johnston ND, Coutre SE, Flinn IW, Schreeder MT, Fowler NH, Sharman JP, Boccia RV, Barrientos JC, Rai KR, Boyd TE, Furman RR, Kim Y, Godfrey WR, Leonard JP. Combinations of idelalisib with rituximab and/or bendamustine in patients with recurrent indolent non-Hodgkin lymphoma. Blood Adv. 2016 Nov 30;1(2):122-131. doi: 10.1182/bloodadvances.2016000976. eCollection 2016 Dec 13. PMID 29296805
- [Derived] Stevenson FK, Krysov S, Davies AJ, Steele AJ, Packham G. B-cell receptor signaling in chronic lymphocytic leukemia. Blood. 2011 Oct 20;118(16):4313-20. doi: 10.1182/blood-2011-06-338855. Epub 2011 Aug 3. PMID 21816833

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States. The first participant was screened on 25 March 2010. The last study visit occurred on 28 April 2015.
Pre-assignment Details: 277 participants were screened. Per prespecified analysis, participants were grouped by disease (chronic lymphocytic leukemia, indolent non-Hodgkin lymphoma, mantle cell lymphoma) and by treatment regimen (cohort).
Groups:
- Idelalisib + Rituximab: Participants with chronic lymphocytic leukemia (CLL) and indolent non-Hodgkin lymphoma (iNHL) received treatments as follows:
  Cohort 1a: Idelalisib (IDELA) 100 mg orally twice daily (BID) on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 intravenously (IV) on Days 1, 8, 15 & 22, Cycles 1 & 2
  Cohort 2a: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Days 1, 8, 15, & 22, Cycles 1 & 2
  Cohort 3e: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Days 1, 8, 15, & 22, Cycles 1 & 2
  Cohort 4a: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle, starting Cycle 2 Day 1 with the 5th dose of rituximab + rituximab 375 mg/m^2 IV on Days 1, 8, 15, & 22, Cycles 1 & 2
- Idelalisib + Bendamustine: Participants with CLL and iNHL received treatments as follows:
  Cohort 1b: IDELA 100 mg orally BID on Days 1 - 28 of each 28-day cycle + bendamustine 90 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
  Cohort 2b: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + bendamustine 90 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
  Cohort 3f: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + bendamustine 90 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
  Cohort 3g: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + bendamustine 70 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
  Cohort 4b: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle starting Cycle 2, Day 3 (after the Cycle 2 bendamustine dosing) + bendamustine 90 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
- Idelalisib + Everolimus: Participants with mantle cell lymphoma (MCL) received treatments as follows:
  Cohort 5a: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + everolimus 10 mg orally once daily on Days 1 - 28 of each 28-day cycle
- Idelalisib + Bortezomib: Participants with MCL received treatments as follows:
  Cohort 5b: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + bortezomib 1.3 mg/m^2 subcutaneously on Days 1, 8 & 15 of each 28-day cycle
- Idelalisib + Rituximab + Bendamustine: Participants with CLL, iNHL and MCL received treatments as follows:
  Cohort 3a: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Day 1 of each 28-day cycle, Cycles 1 - 6 + bendamustine 90 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
  Cohort 3b: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Day 1 of each 28-day cycle, Cycles 1 - 6 + bendamustine 70 mg/m^2 IV on Days 1 & 2 of each 28-day cycle from Cycles 1 - 6
  Cohort 5c: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Day 1 of each 28-day cycle, Cycles 1 - 6 + bendamustine 90 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
- Idelalisib + Ofatumumab: Participants with CLL received treatments as follows:
  Cohort 3c: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + ofatumumab 12 doses (300 mg (Day 1 or Day 2, Dose 1), followed 1 week later by 1,000 mg weekly for 7 doses (Doses 2 - 8), followed 5 weeks later by 1,000 mg every 4 weeks for 4 doses (Doses 9 - 12))
- Idelalisib + Fludarabine: Participants with CLL received treatments as follows:
  Cohort 3d: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + fludarabine 40 mg/m^2 orally on Days 1 - 5 of each 28-day cycle, Cycles 1 - 6
- Idelalisib + Chlorambucil: Participants with CLL received treatments as follows:
  Cohort 6a: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + chlorambucil 10 mg/m^2 orally once daily for 7 days every 28 days, Cycles 1 - 12
- Idelalisib + Rituximab + Chlorambucil: Participants with CLL received treatments as follows:
  Cohort 6b: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Day 1 of each 28-day cycle, Cycles 1 - 6 + chlorambucil 10 mg/m^2 orally once daily for 7 days every 28 days, Cycles 1 - 12
- Idelalisib + Rituximab + Lenalidomide: Participants with CLL and iNHL received treatments as follows:
  Cohort 7a: IDELA 150 mg orally BID on Days 1 - 35 of Cycle 1 (35 days) and Days 1 - 28 of all subsequent 28-day cycles + rituximab 375 mg/m^2 IV on Days 1 & 8 of the first cycle and Day 1 of Cycles 2 - 6 + lenalidomide 5 mg orally once daily starting on Days 8 - 28 of Cycle 1 (35 days) and Days 1 - 21 of the next five 28-day cycles
  Cohort 7b: IDELA 150 mg orally BID on Days 1 - 35 of Cycle 1 (35 days) and Days 1 - 28 of all subsequent 28-day cycles + rituximab 375 mg/m^2 IV on Days 1 & 8 of the first cycle and Day 1 of Cycles 2 - 6 + lenalidomide 10 mg orally once daily starting on Days 8 - 28 of Cycle 1 (35 days) and Days 1 - 21 of the next five 28-day cycles
  Cohort 7c: IDELA 150 mg orally BID on Days 1 - 35 of Cycle 1 (35 days) and Days 1 - 28 of all subsequent 28-day cycles + rituximab 375 mg/m^2 IV on Days 1 & 8 of the first cycle and Day 1 of Cycles 2 - 6 + lenalidomide 20 mg orally once daily starting on Days 8 - 28 of Cycle 1 (35 days) and Days 1 - 21 of the next five 28-day cycles
Period: Overall Study
Arm/Group | Idelalisib + Rituximab | Idelalisib + Bendamustine | Idelalisib + Everolimus | Idelalisib + Bortezomib | Idelalisib + Rituximab + Bendamustine | Idelalisib + Ofatumumab | Idelalisib + Fludarabine | Idelalisib + Chlorambucil | Idelalisib + Rituximab + Chlorambucil | Idelalisib + Rituximab + Lenalidomide
Started | 51 | 51 | 18 | 18 | 33 | 21 | 12 | 15 | 15 | 7
Participants With CLL | 19 | 18 | 0 | 0 | 15 | 21 | 12 | 15 | 14 | 1
Participants With Indolent NHL | 32 | 33 | 0 | 0 | 14 | 0 | 0 | 0 | 1 | 6
Participants With MCL | 0 | 0 | 18 | 18 | 4 | 0 | 0 | 0 | 0 | 0
Completed | 29 | 24 | 4 | 4 | 16 | 10 | 6 | 10 | 8 | 3
Not Completed | 22 | 27 | 14 | 14 | 17 | 11 | 6 | 5 | 7 | 4
Not completed — Adverse Event | 7 | 9 | 7 | 5 | 6 | 3 | 3 | 0 | 2 | 2
Not completed — Withdrew Consent | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 2 | 2 | 1
Not completed — Concomitant Medication Prohibited | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator Request | 2 | 2 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 0
Not completed — Patient Non-compliance | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 7 | 4 | 3 | 5 | 3 | 3 | 2 | 1 | 0 | 0
Not completed — Death | 1 | 5 | 3 | 3 | 1 | 3 | 0 | 0 | 3 | 1
Not completed — Other | 3 | 5 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set included participants who received at least 1 dose of study drug (Idelalisib or combination drugs). Per prespecified analysis, participants were grouped by disease (CLL, iNHL, MCL) and by treatment regimen (cohort).
Groups:
- Idelalisib + Rituximab: Participants with CLL and iNHL received treatments as follows:
  Cohort 1a: IDELA 100 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Days 1, 8, 15 & 22, Cycles 1 & 2
  Cohort 2a: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Days 1, 8, 15, & 22, Cycles 1 & 2
  Cohort 3e: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Days 1, 8, 15, & 22, Cycles 1 & 2
  Cohort 4a: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle, starting Cycle 2 Day 1 with the 5th dose of rituximab + rituximab 375 mg/m^2 IV on Days 1, 8, 15, & 22, Cycles 1 & 2
- Idelalisib + Everolimus: Participants with MCL received treatments as follows:
  Cohort 5a: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + everolimus 10 mg orally once daily on Days 1 - 28 of each 28-day cycle
- Total: Total of all reporting groups
Arm/Group | Idelalisib + Rituximab | Idelalisib + Bendamustine | Idelalisib + Everolimus | Idelalisib + Bortezomib | Idelalisib + Rituximab + Bendamustine | Idelalisib + Ofatumumab | Idelalisib + Fludarabine | Idelalisib + Chlorambucil | Idelalisib + Rituximab + Chlorambucil | Idelalisib + Rituximab + Lenalidomide | Total
Number analyzed (Participants) | 51 | 51 | 18 | 18 | 33 | 21 | 12 | 15 | 15 | 7 | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (10.1) | 61 (11.2) | 69 (7.1) | 72 (6.0) | 60 (8.3) | 66 (9.7) | 69 (7.1) | 63 (7.8) | 68 (10.0) | 61 (8.3) | 64 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 21 | 7 | 3 | 12 | 6 | 4 | 1 | 4 | 2 | 76
  Male | 35 | 30 | 11 | 15 | 21 | 15 | 8 | 14 | 11 | 5 | 165
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 42 | 45 | 16 | 14 | 29 | 20 | 8 | 14 | 15 | 6 | 209
  Black or African American | 2 | 3 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 9
  Asian | 5 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 11
  Other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Not Reported | 2 | 2 | 1 | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 4
  Not Hispanic or Latino | 51 | 49 | 18 | 17 | 31 | 21 | 11 | 14 | 15 | 7 | 234
  Missing | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Duration of Exposure to IDELA
Description: Duration of exposure to IDELA was summarized using descriptive statistics.
Time Frame: First dose date up to 12 months
Population: The ITT analysis set included participants who received at least 1 dose of study drug (idelalisib or combination drugs). Per prespecified analysis, participants for this outcome measure were grouped by disease and treatment regimen (cohort).
Measure: Mean (Standard Deviation); unit: months
Groups:
- Idelalisib + Rituximab: Participants with chronic CLL and iNHL received treatments as follows:
  Cohort 1a: IDELA 100 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Days 1, 8, 15 & 22, Cycles 1 & 2
  Cohort 2a: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Days 1, 8, 15, & 22, Cycles 1 & 2
  Cohort 3e: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Days 1, 8, 15, & 22, Cycles 1 & 2
  Cohort 4a: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle, starting Cycle 2 Day 1 with the 5th dose of rituximab + rituximab 375 mg/m^2 IV on Days 1, 8, 15, & 22, Cycles 1 & 2
Arm/Group | Idelalisib + Rituximab | Idelalisib + Bendamustine | Idelalisib + Everolimus | Idelalisib + Bortezomib | Idelalisib + Rituximab + Bendamustine | Idelalisib + Ofatumumab | Idelalisib + Fludarabine | Idelalisib + Chlorambucil | Idelalisib + Rituximab + Chlorambucil | Idelalisib + Rituximab + Lenalidomide
Number analyzed (Participants) | 51 | 51 | 18 | 18 | 33 | 21 | 12 | 15 | 15 | 7
months | 8.1 (3.74) | 7.6 (3.96) | 4.2 (3.92) | 5.1 (3.90) | 8.0 (4.16) | 8.3 (4.03) | 8.9 (3.57) | 8.8 (3.76) | 8.7 (3.01) | 7.7 (4.78)

2. Primary Outcome: Toxicity of Administration of IDELA
Description: Percentage of participants experiencing toxicities of administration of IDELA were measured according to the Common Terminology Criteria for Adverse Events v4.02
Time Frame: First dose date up to 5 years
Population: Participants in the ITT analysis set were analyzed. Per prespecified analysis, participants for this outcome measure were grouped by disease and treatment regimen (cohort).
Measure: Number; unit: percentage of participants
Arm/Group | Idelalisib + Rituximab | Idelalisib + Bendamustine | Idelalisib + Everolimus | Idelalisib + Bortezomib | Idelalisib + Rituximab + Bendamustine | Idelalisib + Ofatumumab | Idelalisib + Fludarabine | Idelalisib + Chlorambucil | Idelalisib + Rituximab + Chlorambucil | Idelalisib + Rituximab + Lenalidomide
Number analyzed (Participants) | 51 | 51 | 18 | 18 | 33 | 21 | 12 | 15 | 15 | 7
percentage of participants | 100.0 | 100.0 | 100.0 | 83.33 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

3. Secondary Outcome: Overall Response Rate
Description: Overall Response Rate (ORR) was defined as the percentage of participants achieving a complete response (CR) or partial response (PR).
  The response definitions were based on the following standard criteria established for each indication:
  * CLL: International Workshop on chronic lymphocytic leukemia (IWCLL),2008
  * iNHL & MCL: Cheson, 2007
Time Frame: Up to 5 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Idelalisib + Rituximab | Idelalisib + Bendamustine | Idelalisib + Everolimus | Idelalisib + Bortezomib | Idelalisib + Rituximab + Bendamustine | Idelalisib + Ofatumumab | Idelalisib + Fludarabine | Idelalisib + Chlorambucil | Idelalisib + Rituximab + Chlorambucil | Idelalisib + Rituximab + Lenalidomide
Number analyzed (Participants) | 51 | 51 | 18 | 18 | 33 | 21 | 12 | 15 | 15 | 7
percentage of participants | 78.4 [64.7 to 88.7] | 84.3 [71.4 to 93.0] | 44.4 [21.5 to 69.2] | 61.1 [35.7 to 82.7] | 81.8 [64.5 to 93.0] | 71.4 [47.8 to 88.7] | 91.7 [61.5 to 99.8] | 66.7 [38.4 to 88.2] | 93.3 [68.1 to 99.8] | 71.4 [29.0 to 96.3]

4. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) was defined as the interval from the first documentation of CR or PR to the earlier of the first documentation of disease progression or death from any cause.
Time Frame: Up to 5 years
Population: Participants in the ITT analysis set with available data were analyzed. Per prespecified analysis, participants for this outcome measure were grouped by disease and treatment regimen (cohort).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Idelalisib + Rituximab | Idelalisib + Bendamustine | Idelalisib + Everolimus | Idelalisib + Bortezomib | Idelalisib + Rituximab + Bendamustine | Idelalisib + Ofatumumab | Idelalisib + Fludarabine | Idelalisib + Chlorambucil | Idelalisib + Rituximab + Chlorambucil | Idelalisib + Rituximab + Lenalidomide
Number analyzed (Participants) | 40 | 43 | 8 | 11 | 27 | 15 | 11 | 10 | 14 | 5
months | NA [NA to NA] — NA = Not Reached; too few events to estimate the median and the lower and upper limits of the confidence interval | NA [NA to NA] — NA = Not Reached; too few events to estimate the median and the lower and upper limits of the confidence interval | 5.6 [1.1 to NA] — NA = Not Reached; too few events to estimate the upper limit of the confidence interval | 9.3 [4.9 to 9.3] | NA [9.9 to NA] — NA = Not Reached; too few events to estimate the median and the upper limit of the confidence interval | NA [9.4 to NA] — NA = Not Reached; too few events to estimate the median and the upper limit of the confidence interval | NA [3.5 to NA] — NA = Not Reached; too few events to estimate the median and the upper limit of the confidence interval | NA [NA to NA] — NA = Not Reached; too few events to estimate the median and the lower and upper limits of the confidence interval | NA [4.4 to NA] — NA = Not Reached; too few events to estimate the median and the upper limit of the confidence interval | NA [1.3 to NA] — NA = Not Reached; too few events to estimate the median and the upper limit of the confidence interval

5. Secondary Outcome: Time to Response
Description: Time to response (TTR) was defined as the interval from the start of study drug to the first documentation of CR or PR.
Time Frame: Up to 5 years
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Idelalisib + Rituximab | Idelalisib + Bendamustine | Idelalisib + Everolimus | Idelalisib + Bortezomib | Idelalisib + Rituximab + Bendamustine | Idelalisib + Ofatumumab | Idelalisib + Fludarabine | Idelalisib + Chlorambucil | Idelalisib + Rituximab + Chlorambucil | Idelalisib + Rituximab + Lenalidomide
Number analyzed (Participants) | 40 | 43 | 8 | 11 | 27 | 15 | 11 | 10 | 14 | 5
months | 1.9 [1.9 to 2.1] | 1.9 [1.9 to 2.0] | 1.9 [1.9 to 2.6] | 1.9 [1.9 to 1.9] | 1.9 [1.9 to 2.0] | 1.9 [1.9 to 2.3] | 1.9 [1.8 to 1.9] | 1.9 [1.9 to 1.9] | 1.9 [1.9 to 3.7] | 3.0 [2.6 to 4.0]

6. Secondary Outcome: Progression-free Survival
Description: Progression free survival (PFS) was defined as the interval from the start of study drug to the earlier of the first documentation of disease progression or death from any cause.
  The response definitions were based on the following standard criteria established for each indication:
  * CLL: International Workshop on chronic lymphocytic leukemia (IWCLL), 2008
  * iNHL & MCL: Cheson, 2007
Time Frame: Up to 5 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Idelalisib + Rituximab | Idelalisib + Bendamustine | Idelalisib + Everolimus | Idelalisib + Bortezomib | Idelalisib + Rituximab + Bendamustine | Idelalisib + Ofatumumab | Idelalisib + Fludarabine | Idelalisib + Chlorambucil | Idelalisib + Rituximab + Chlorambucil | Idelalisib + Rituximab + Lenalidomide
Number analyzed (Participants) | 51 | 51 | 18 | 18 | 33 | 21 | 12 | 15 | 15 | 7
months | NA [NA to NA] — NA = Not Reached; too few events to estimate the median and the lower and upper limits of the confidence interval | NA [NA to NA] — NA = Not Reached; too few events to estimate the median and the lower and upper limits of the confidence interval | 4.3 [1.6 to 11.1] | 8.1 [1.8 to NA] — NA = Not Reached; too few events to estimate the upper limit of the confidence interval | NA [11.7 to NA] — NA = Not Reached; too few events to estimate the median and the upper limit of the confidence interval | NA [8.7 to NA] — NA = Not Reached; too few events to estimate the median and the upper limit of the confidence interval | NA [5.4 to NA] — NA = Not Reached; too few events to estimate the median and the upper limit of the confidence interval | NA [NA to NA] — NA = Not Reached; too few events to estimate the median and the lower and upper limits of the confidence interval | NA [6.7 to NA] — NA = Not Reached; too few events to estimate the median and the upper limit of the confidence interval | NA [5.5 to NA] — NA = Not Reached; too few events to estimate the median and the upper limit of the confidence interval

7. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) was defined as the interval from the start of study drug to death from any cause.
Time Frame: Up to 5 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Idelalisib + Rituximab | Idelalisib + Bendamustine | Idelalisib + Everolimus | Idelalisib + Bortezomib | Idelalisib + Rituximab + Bendamustine | Idelalisib + Ofatumumab | Idelalisib + Fludarabine | Idelalisib + Chlorambucil | Idelalisib + Rituximab + Chlorambucil | Idelalisib + Rituximab + Lenalidomide
Number analyzed (Participants) | 51 | 51 | 18 | 18 | 33 | 21 | 12 | 15 | 15 | 7
months | NA [NA to NA] — NA = Not Reached; too few events to estimate the median and the lower and upper limits of the confidence interval | NA [NA to NA] — NA = Not Reached; too few events to estimate the median and the lower and upper limits of the confidence interval | NA [3.4 to NA] — NA = Not Reached; too few events to estimate the median and the upper limit of the confidence interval | NA [5.2 to NA] — NA = Not Reached; too few events to estimate the median and the upper limit of the confidence interval | NA [NA to NA] — NA = Not Reached; too few events to estimate the median and the lower and upper limits of the confidence interval | NA [NA to NA] — NA = Not Reached; too few events to estimate the median and the lower and upper limits of the confidence interval | NA [6.3 to NA] — NA = Not Reached; too few events to estimate the median and the upper limit of the confidence interval | NA [NA to NA] — NA = Not Reached; too few events to estimate the median and the lower and upper limits of the confidence interval | NA [6.7 to NA] — NA = Not Reached; too few events to estimate the median and the upper limit of the confidence interval | NA [5.5 to NA] — NA = Not Reached; too few events to estimate the median and the upper limit of the confidence interval

8. Secondary Outcome: Plasma Concentration of IDELA (Cohort 1, Cohorts 2 and 3, Cohort 5)
Time Frame: Predose, 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0 hours postdose at Week 0; predose, 1.5 hours postdose at Weeks 4, 12, and 24
Population: The pharmacokinetic (PK) analysis set included data from participants in the ITT analysis set who had the necessary baseline and on-study measurements to provide interpretable results for the specific parameters of interest. Per prespecified analysis, data were summarized for participants in Cohort 1a 1b, who received idelalisib 100 mg and for participants in Cohorts 2a, 2b, 3a, 3b, 3c, 3d, 3e, 3f, 3g 5a, 5b, and 5c who received idelalisib 150 mg.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Idelalisib 100 mg (Cohort 1): Participants analyzed for this group included participants from Cohort 1 (subcohort 1a and 1b) who received the treatments as follows:
  Cohort 1a: IDELA 100 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Days 1, 8, 15 & 22, Cycles 1 & 2
  Cohort 1b: IDELA 100 mg orally BID on Days 1 - 28 of each 28-day cycle + bendamustine 90 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycle 1 - 6
- Idelalisib 150 mg (Cohorts 2 and 3): Participants analyzed for this group included participants from Cohort 2a, 2b, 3a, 3b, 3c, 3e, 3f, 3g who received the treatments as follows:
  Cohort 2a: IDELA 150 mg orally (po) BID, D1 - D28 of each cycle + rituximab 375 mg/m^2 IV on D1, D8, D15, & D22, C1 & C2
  Cohort 2b: IDELA 150 mg po BID, D1 - D28 of each cycle + bendamustine 90 mg/m^2 IV, D1 & D2, C1 - C6
  Cohorts 3a and 3b: IDELA 150 mg po BID, D1 - D28 of each cycle + rituximab 375 mg/m^2 IV on D1, C1 - C6 + bendamustine 90 mg/m^2 (Cohort 3a only) IV, D1 & D2, C1 - C6 + bendamustine 70 mg/m^2 (Cohort 3b only) IV on D1 & D2, C1 - C6
  Cohort 3c: IDELA 150 mg po BID, D1 - D28 of each cycle + ofatumumab 12 doses (300 mg (D1 or D2, Dose 1), followed 1 week later by 1,000 mg weekly for 7 doses (Doses 2 - 8), followed 5 weeks later by 1,000 mg every 4 weeks for 4 doses (Doses 9 - 12))
  Cohort 3d: IDELA 150 mg po BID, D1 - D28 of each cycle + fludarabine 40 mg/m^2 po D1 - D5, C1 - C6
  Cohort 3e: IDELA 150 mg po BID, D1 - D28 of each cycle + rituximab 375 mg/m^2 IV on D1, D8, D15, & D22, C1 & C2
  Cohorts 3f and 3g: IDELA 150 mg po BID, D1 - D28 of each cycle + bendamustine 90 mg/m^2 (cohort 3f only) IV, D1 & D2, C1 - C6 + bendamustine 70 mg/m^2 (Cohort 3g only) IV, D1 & D2, C1 - C6
  C= Cycle D= Day Cycle length= 28 days
- Idelalisib 150 mg (Cohort 5): Participants analyzed for this group included participants from Cohort 5 (subcohorts 5a, 5b, and 5c) who received the treatments as follows:
  Cohort 5a: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + everolimus 10 mg orally once daily on Days 1 - 28 of each 28-day cycle
  Cohort 5b: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + bortezomib 1.3 mg/m^2 subcutaneously on Days 1, 8 & 15 of each 28-day cycle
  Cohort 5c: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Day 1 of each 28-day cycle, Cycles 1 - 6 + bendamustine 90 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
Arm/Group | Idelalisib 100 mg (Cohort 1) | Idelalisib 150 mg (Cohorts 2 and 3) | Idelalisib 150 mg (Cohort 5)
Number analyzed (Participants) | 24 | 123 | 45
ng/mL
  Pre-dose (Week 0): number analyzed (Participants) | 24 | 111 | 36
  Pre-dose (Week 0) | 0.4 (2.16) | 68.8 (396.94) | 0.0 (0.0)
  0.5 hr post-dose (Week 0): number analyzed (Participants) | 7 | 22 | 1
  0.5 hr post-dose (Week 0) | 437.6 (380.08) | 1231.4 (1238.20) | 1380.0
  1.0 hr post-dose (Week 0): number analyzed (Participants) | 7 | 22 | 1
  1.0 hr post-dose (Week 0) | 1022.4 (652.92) | 1789.3 (1162.31) | 1600.0
  1.5 hr post-dose (Week 0): number analyzed (Participants) | 24 | 112 | 36
  1.5 hr post-dose (Week 0) | 1434.0 (835.25) | 2017.3 (1241.96) | 1564.7 (983.46)
  2.0 hr post-dose (Week 0): number analyzed (Participants) | 7 | 21 | 1
  2.0 hr post-dose (Week 0) | 1282.7 (789.24) | 1732.8 (744.87) | 1400.0
  3.0 hr post-dose (Week 0): number analyzed (Participants) | 7 | 22 | 1
  3.0 hr post-dose (Week 0) | 1001.0 (633.99) | 1296.1 (509.80) | 1170.0
  4.0 hr post-dose (Week 0): number analyzed (Participants) | 7 | 22 | 1
  4.0 hr post-dose (Week 0) | 788.4 (629.67) | 910.0 (420.79) | 795.0
  6.0 hr post-dose (Week 0): number analyzed (Participants) | 7 | 21 | 1
  6.0 hr post-dose (Week 0) | 523.7 (418.80) | 486.0 (276.75) | 517.0
  Pre-dose (Week 4): number analyzed (Participants) | 22 | 99 | 29
  Pre-dose (Week 4) | 416.5 (636.01) | 364.1 (341.84) | 408.0 (699.35)
  1.5 hr post-dose (Week 4): number analyzed (Participants) | 20 | 95 | 24
  1.5 hr post-dose (Week 4) | 1297.2 (681.43) | 1808.1 (931.67) | 1877.9 (859.74)
  Pre-dose (Week 12): number analyzed (Participants) | 19 | 78 | 16
  Pre-dose (Week 12) | 361.9 (580.70) | 351.4 (389.78) | 433.9 (529.79)
  1.5 hr post-dose (Week 12): number analyzed (Participants) | 17 | 77 | 12
  1.5 hr post-dose (Week 12) | 1309.5 (750.50) | 1883.0 (973.26) | 1426.8 (917.02)
  Pre-dose (Week 24): number analyzed (Participants) | 11 | 76 | 7
  Pre-dose (Week 24) | 369.9 (461.67) | 419.7 (359.03) | 549.1 (622.95)
  1.5 hr post-dose (Week 24): number analyzed (Participants) | 8 | 72 | 5
  1.5 hr post-dose (Week 24) | 1061.6 (567.90) | 1840.1 (1035.91) | 885.6 (568.81)

9. Secondary Outcome: Plasma Concentration of IDELA (Cohort 4)
Time Frame: Predose at Week 0; predose, 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0 hours postdose at Week 4; predose, 1.5 hours postdose at Week 12; and predose, 1.5 hours postdose at Week 24
Population: Participants in the PK analysis set with available data were analyzed. Per prespecified analysis, data were summarized for participants in Cohort 4a, 4b who received idelalisib 150mg.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Idelalisib 150 mg (Cohort 4): Participants analyzed for this group included participants from Cohort 4 (subcohorts 4a and 4b) who received the treatments as follows:
  Cohort 4a: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle, starting Cycle 2 Day 1 with the 5th dose of rituximab + rituximab 375 mg/m^2 IV on Days 1, 8, 15, & 22, Cycles 1 & 2
  Cohort 4b: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle starting Cycle 2, Day 3 (after the Cycle 2 bendamustine dosing) + bendamustine 90 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
Arm/Group | Idelalisib 150 mg (Cohort 4)
Number analyzed (Participants) | 18
ng/mL
  Pre-dose (Week 0): number analyzed (Participants) | 3
  Pre-dose (Week 0) | 0.0 (0.0)
  Pre-dose (Week 4): number analyzed (Participants) | 13
  Pre-dose (Week 4) | 0.0 (0.0)
  0.5 hr post-dose (Week 4): number analyzed (Participants) | 2
  0.5 hr post-dose (Week 4) | 1119.5 (1513.99)
  1.0 hr post-dose (Week 4): number analyzed (Participants) | 2
  1.0 hr post-dose (Week 4) | 994.5 (601.75)
  1.5 hr post-dose (Week 4): number analyzed (Participants) | 12
  1.5 hr post-dose (Week 4) | 1758.2 (1414.07)
  2.0 hr post-dose (Week 4): number analyzed (Participants) | 2
  2.0 hr post-dose (Week 4) | 737.0 (108.89)
  3.0 hr post-dose (Week 4): number analyzed (Participants) | 2
  3.0 hr post-dose (Week 4) | 605.0 (18.38)
  4.0 hr post-dose (Week 4): number analyzed (Participants) | 2
  4.0 hr post-dose (Week 4) | 547.0 (158.39)
  6.0 hr post-dose (Week 4): number analyzed (Participants) | 2
  6.0 hr post-dose (Week 4) | 524.0 (404.47)
  Pre-dose (Week 12): number analyzed (Participants) | 13
  Pre-dose (Week 12) | 401.9 (344.93)
  1.5 hr post-dose (Week 12): number analyzed (Participants) | 11
  1.5 hr post-dose (Week 12) | 2018.2 (1703.98)
  Pre-dose (Week 24): number analyzed (Participants) | 12
  Pre-dose (Week 24) | 752.5 (967.91)
  1.5 hr post-dose (Week 24): number analyzed (Participants) | 10
  1.5 hr post-dose (Week 24) | 2251.1 (1744.44)

10. Secondary Outcome: Plasma Concentration of IDELA (Cohort 6)
Time Frame: Predose, 1.5 hours postdose at Weeks 0, 4, 12 and 24
Population: Participants in the PK analysis set with available data were analyzed. Per prespecified analysis, data were summarized for participants in Cohort 6a, 6b who received idelalisib 150mg.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Idelalisib 150 mg (Cohort 6): Participants analyzed for this group included participants from Cohort 6 (subcohorts 6a and 6b) who received the treatments as follows
  Cohort 6a: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + chlorambucil 10 mg/m^2 orally once daily for 7 days every 28 days, Cycles 1 - 12
  Cohort 6b: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Day 1 of each 28-day cycle, Cycles 1 - 6 + chlorambucil 10 mg/m^2 orally once daily for 7 days every 28 days, Cycles 1 - 12
Arm/Group | Idelalisib 150 mg (Cohort 6)
Number analyzed (Participants) | 30
ng/mL
  Pre-dose (Week 0) | 0.0 (0.0)
  1.5 hr post-dose (Week 0): number analyzed (Participants) | 27
  1.5 hr post-dose (Week 0) | 1930.7 (1220.87)
  Pre-dose (Week 4): number analyzed (Participants) | 24
  Pre-dose (Week 4) | 530.8 (563.59)
  1.5 hr post-dose (Week 4): number analyzed (Participants) | 22
  1.5 hr post-dose (Week 4) | 1869.8 (1001.39)
  Pre-dose (Week 12): number analyzed (Participants) | 25
  Pre-dose (Week 12) | 677.9 (940.94)
  1.5 hr post-dose (Week 12): number analyzed (Participants) | 18
  1.5 hr post-dose (Week 12) | 1733.0 (941.94)
  Pre-dose (Week 24): number analyzed (Participants) | 21
  Pre-dose (Week 24) | 346.8 (377.84)
  1.5 hr post-dose (Week 24): number analyzed (Participants) | 19
  1.5 hr post-dose (Week 24) | 1710.7 (1235.08)

11. Secondary Outcome: Plasma Concentration of IDELA (Cohort 7)
Time Frame: Predose, 1.5 hours postdose at Weeks 0, 5 and 13
Population: Participants in the PK analysis set with available data were analyzed. Per prespecified analysis, data were summarized for participants in Cohort 7a, 7b, 7c who received idelalisib 150mg.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Idelalisib 150 mg (Cohort 7): Participants analyzed for this group included participants from Cohort 7 (subcohorts 7a, 7b, and 7c) who received the treatments as follows:
  Cohort 7a: IDELA 150 mg orally BID on Days 1 - 35 of Cycle 1 (35 days) and Days 1 - 28 of all subsequent 28-day cycles + rituximab 375 mg/m^2 IV on Days 1 & 8 of the first cycle and Day 1 of Cycles 2 - 6 + lenalidomide 5 mg orally once daily starting on Days 8 - 28 of Cycle 1 (35 days) and Days 1 - 21 of the next five 28-day cycles
  Cohort 7b: IDELA 150 mg orally BID on Days 1 - 35 of Cycle 1 (35 days) and Days 1 - 28 of all subsequent 28-day cycles + rituximab 375 mg/m^2 IV on Days 1 & 8 of the first cycle and Day 1 of Cycles 2 - 6 + lenalidomide 10 mg orally once daily starting on Days 8 - 28 of Cycle 1 (35 days) and Days 1 - 21 of the next five 28-day cycles
  Cohort 7c: IDELA 150 mg orally BID on Days 1 - 35 of Cycle 1 (35 days) and Days 1 - 28 of all subsequent 28-day cycles + rituximab 375 mg/m^2 IV on Days 1 & 8 of the first cycle and Day 1 of Cycles 2 - 6 + lenalidomide 20 mg orally once daily starting on Days 8 - 28 of Cycle 1 (35 days) and Days 1 - 21 of the next five 28-day cycles
Arm/Group | Idelalisib 150 mg (Cohort 7)
Number analyzed (Participants) | 7
ng/mL
  Pre-dose (Week 0) | NA (NA) — Values were below the limit of quantitation
  1.5 hr post-dose (Week 0) | 1603.1 (1196.78)
  Pre-dose (Week 5): number analyzed (Participants) | 6
  Pre-dose (Week 5) | 20.7 (50.13)
  1.5 hr post-dose (Week 5): number analyzed (Participants) | 6
  1.5 hr post-dose (Week 5) | 1621.3 (663.80)
  Pre-dose (Week 13): number analyzed (Participants) | 4
  Pre-dose (Week 13) | 354.8 (278.62)
  1.5 hr post-dose (Week 13): number analyzed (Participants) | 3
  1.5 hr post-dose (Week 13) | 592.7 (597.52)

12. Secondary Outcome: Sub-study: Plasma Concentration of IDELA (Cohorts 1-4)
Time Frame: pre dose and 0.5, 1, 1.5, 2.0, 3.0, 4.0, and 6.0 hours post dose
Population: Participants with CLL or iNHL from the PK Analysis Set in Cohorts 1, 2, 3, and 4 who participated in the PK substudy were analyzed. Per prespecified analysis, data were summarized for participants in Cohort 1a, 1b who received idelalisib 100mg and Cohorts 2a, 2b, 3a, 3c, 3d, 3e, 3f, 3g, 4a, 4b who received idelalisib 150 mg in the PK substudy.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Idelalisib 100 mg (Cohort 1a, 1b): Participants analyzed for this group included participants from Cohort 1 who received the treatments as follows:
  Cohort 1a: IDELA 100 mg orally BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Days 1, 8, 15 & 22, Cycles 1 & 2
  Cohort 1b: IDELA 100 mg orally BID on Days 1 - 28 of each 28-day cycle + bendamustine 90 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
- Idelalisib 150 mg (Cohorts 2a, 2b, 3a, 3c, 3d, 3e, 3f, 3g, 4a, 4b): Participants included for analysis received treatments as follows:
  Cohort 2a: IDELA 150 mg po BID, D1 - D28 of each cycle + rituximab 375 mg/m^2 IV on D1, D8, D15, & D22, C1 & C2
  Cohort 2b: IDELA 150 mg po BID, D1 - D28 of each cycle + bendamustine 90 mg/m^2 IV, D1 & D2, C1 - C6
  Cohorts 3a and 3b: IDELA 150 mg po BID, D1 - D28 of each cycle + rituximab 375 mg/m^2 IV on D1, C1 - C6 + bendamustine 90 mg/m^2 (Cohort 3a only) IV, D1 & D2, C1 - C6 + bendamustine 70 mg/m^2 (Cohort 3b only) IV on D1 & D2, C1 - C6
  Cohort 3c: IDELA 150 mg po BID, D1 - D28 of each cycle + ofatumumab 12 doses (300 mg (D1 or D2, Dose 1), followed 1 week later by 1,000 mg weekly for 7 doses (Doses 2 - 8), followed 5 weeks later by 1,000 mg every 4 weeks for 4 doses (Doses 9 - 12))
  Cohort 3d: IDELA 150 mg po BID, D1 - D28 of each cycle + fludarabine 40 mg/m^2 po D1 - D5, C1 - C6
  Cohort 3e: IDELA 150 mg po BID, D1 - D28 of each cycle + rituximab 375 mg/m^2 IV on D1, D8, D15, & D22, C1 & C2
  Cohorts 3f and 3g: IDELA 150 mg po BID, D1 - D28 of each cycle + bendamustine 90 mg/m^2 (Cohort 3f only) IV, D1 & D2, C1 - C6 + bendamustine 70 mg/m^2 (Cohort 3g only) IV, D1 & D2, C1 - C6
  Cohort 4a: IDELA 150 mg po BID, D1 - D28 of each cycle (starting C2 D1) + rituximab 375 mg/m^2 IV, D1, D8, D15, & D22, C1 & C2
  Cohort 4b: IDELA 150 mg po BID, D1 - D28 of each cycle (starting C2, D3) + bendamustine 90 mg/m^2 IV, D1 & D2, C1 - C6
  C= Cycle D= Day Cycle length= 28 days
Arm/Group | Idelalisib 100 mg (Cohort 1a, 1b) | Idelalisib 150 mg (Cohorts 2a, 2b, 3a, 3c, 3d, 3e, 3f, 3g, 4a, 4b)
Number analyzed (Participants) | 7 | 24
ng/mL
  Pre-dose | 1.5 (4.01) | 0.0 (0.0)
  0.5 hr post-dose | 437.6 (380.08) | 1222.1 (1224.95)
  1.0 hr post-dose | 1022.4 (652.92) | 1723.1 (1140.00)
  1.5 hr post-dose | 1264.7 (868.41) | 1599.2 (746.58)
  2.0 hr post-dose: number analyzed (Participants) | 7 | 23
  2.0 hr post-dose | 1282.7 (789.24) | 1646.2 (766.31)
  3.0 hr post-dose | 1001.0 (633.99) | 1238.5 (524.77)
  4.0 hr post-dose | 788.4 (629.67) | 879.8 (416.25)
  6.0 hr post-dose: number analyzed (Participants) | 7 | 23
  6.0 hr post-dose | 523.7 (418.80) | 489.3 (277.82)

13. Secondary Outcome: Plasma Concentration of Bendamustine
Time Frame: Predose, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2.0, 3.0, 4.0, 5.0, 6.0 hours postdose at Week 0
Population: Participants in the PK analysis set with available data were analyzed. Per prespecified analysis, data were summarized for participants in Cohorts 1b, 2b, 3a, 3b, 3f, 3g, 4b, 5c who received bendamustine.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Bendamustine (Cohorts 1b, 2b, 3a, 3b, 3f, 3g, 4b, 5c): Participants included for analysis received treatments as follows:
  Cohort 1b: IDELA 100 mg po BID on Days 1 - 28 of each 28-day cycle + bendamustine 90 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
  Cohort 2b: IDELA 150 mg po BID on Days 1 - 28 of each 28-day cycle + bendamustine 90 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
  Cohort 3a: IDELA 150 mg po BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Day 1 of each 28-day cycle, Cycles 1 - 6 + bendamustine 90 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
  Cohort 3b: IDELA 150 mg po BID on Days 1 - 28 of each 28-day cycle + rituximab 375 mg/m^2 IV on Day 1 of each 28-day cycle, Cycles 1 - 6 + bendamustine 70 mg/m^2 IV on Days 1 & 2 of each 28-day cycle from Cycles 1 - 6
  Cohort 3f: IDELA 150 mg po BID on Days 1 - 28 of each 28-day cycle + bendamustine 90 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
  Cohort 3g: IDELA 150 mg po BID on Days 1 - 28 of each 28-day cycle + bendamustine 70 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
  Cohort 4b: IDELA 150 mg po BID on Days 1 - 28 of each 28-day cycle starting Cycle 2, Day 3 (after the Cycle 2 bendamustine dosing) + bendamustine 90 mg/m^2 IV on Days 1 & 2 of each 28-day cycle, Cycles 1 - 6
  Cohort 5c: IDELA 150 mg po BID on Days 1 - 28 + rituximab 375 mg/m^2 IV on Day 1, Cycles 1 - 6 + bendamustine 90 mg/m^2 IV on Days 1 & 2, Cycles 1 - 6 (Cycle length= 28 days)
Arm/Group | Bendamustine (Cohorts 1b, 2b, 3a, 3b, 3f, 3g, 4b, 5c)
Number analyzed (Participants) | 19
ng/mL
  Pre-dose (Week 0) | NA (NA) — Values were below the limit of quantitation
  0.25 hr post-dose (Week 0): number analyzed (Participants) | 18
  0.25 hr post-dose (Week 0) | 3484.1 (2617.17)
  0.5 hr post-dose (Week 0): number analyzed (Participants) | 18
  0.5 hr post-dose (Week 0) | 4694.7 (3570.78)
  0.75 hr post-dose (Week 0) | 3433.2 (2991.15)
  1.0 hr post-dose (Week 0): number analyzed (Participants) | 18
  1.0 hr post-dose (Week 0) | 2847.2 (2462.90)
  1.25 hr post-dose (Week 0): number analyzed (Participants) | 18
  1.25 hr post-dose (Week 0) | 1916.4 (1551.50)
  1.5 hr post-dose (Week 0): number analyzed (Participants) | 17
  1.5 hr post-dose (Week 0) | 1211.2 (1093.74)
  2.0 hr post-dose (Week 0): number analyzed (Participants) | 18
  2.0 hr post-dose (Week 0) | 514.0 (489.76)
  3.0 hr post-dose (Week 0): number analyzed (Participants) | 18
  3.0 hr post-dose (Week 0) | 463.4 (1529.30)
  4.0 hr post-dose (Week 0): number analyzed (Participants) | 18
  4.0 hr post-dose (Week 0) | 78.5 (238.30)
  5.0 hr post-dose (Week 0): number analyzed (Participants) | 18
  5.0 hr post-dose (Week 0) | 15.3 (36.79)
  6.0 hr post-dose (Week 0): number analyzed (Participants) | 16
  6.0 hr post-dose (Week 0) | 4.4 (6.58)

14. Secondary Outcome: Plasma Concentration of Everolimus
Time Frame: Predose, 1.5 hours postdose at Weeks 0 and 4
Population: Participants in the PK analysis set with available data were analyzed. Data were summarized for participants in Cohort 5a who received everolimus.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Everolimus (Cohort 5a): Participants analyzed for this group included participants from Cohort 5 (subcohort 5a) who received the treatments as follows:
  Cohort 5a: IDELA 150 mg orally BID on Days 1 - 28 of each 28-day cycle + everolimus 10 mg orally once daily on Days 1 - 28 of each 28-day cycle
Arm/Group | Everolimus (Cohort 5a)
Number analyzed (Participants) | 6
ng/mL
  Pre-dose (Week 0): number analyzed (Participants) | 4
  Pre-dose (Week 0) | NA (NA) — Values were below the limit of quantitation
  1.5 hr post-dose (Week 0) | 93.0 (63.50)
  Pre-dose (Week 4): number analyzed (Participants) | 2
  Pre-dose (Week 4) | 3.0 (3.79)
  1.5 hr post-dose (Week 4): number analyzed (Participants) | 2
  1.5 hr post-dose (Week 4) | 56.3 (67.48)

15. Secondary Outcome: Plasma Concentration of Lenalidomide
Time Frame: Predose, 1.5 hours postdose at Week 1 and predose at Week 5
Population: Participants in the PK analysis set with available data were analyzed. Per prespecified analysis, data were summarized for participants in Cohort 7a, 7b, 7c who received lenalidomide.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Lenalidomide (Cohort 7a, 7b, 7c): Participants analyzed for this group included participants from Cohort 7 (subcohorts 7a, 7b, and 7c) who received the treatments as follows:
  Cohort 7a: IDELA 150 mg orally BID on Days 1 - 35 of Cycle 1 (35 days) and Days 1 - 28 of all subsequent 28-day cycles + rituximab 375 mg/m^2 IV on Days 1 & 8 of the first cycle and Day 1 of Cycles 2 - 6 + lenalidomide 5 mg orally once daily starting on Days 8 - 28 of Cycle 1 (35 days) and Days 1 - 21 of the next five 28-day cycles
  Cohort 7b: IDELA 150 mg orally BID on Days 1 - 35 of Cycle 1 (35 days) and Days 1 - 28 of all subsequent 28-day cycles + rituximab 375 mg/m^2 IV on Days 1 & 8 of the first cycle and Day 1 of Cycles 2 - 6 + lenalidomide 10 mg orally once daily starting on Days 8 - 28 of Cycle 1 (35 days) and Days 1 - 21 of the next five 28-day cycles
  Cohort 7c: IDELA 150 mg orally BID on Days 1 - 35 of Cycle 1 (35 days) and Days 1 - 28 of all subsequent 28-day cycles + rituximab 375 mg/m^2 IV on Days 1 & 8 of the first cycle and Day 1 of Cycles 2 - 6 + lenalidomide 20 mg orally once daily starting on Days 8 - 28 of Cycle 1 (35 days) and Days 1 - 21 of the next five 28-day cycles
Arm/Group | Lenalidomide (Cohort 7a, 7b, 7c)
Number analyzed (Participants) | 7
ng/mL
  Pre-dose (Week 1) | NA (NA) — Values were below the limit of quantitation
  1.5 hr post-dose (Week 1): number analyzed (Participants) | 6
  1.5 hr post-dose (Week 1) | 51.6 (31.77)
  Pre-dose (Week 5): number analyzed (Participants) | 2
  Pre-dose (Week 5) | NA (NA) — Values were below the limit of quantitation

ADVERSE EVENTS:
Time Frame: First dose date up to 5 years
Description: The ITT analysis set included participants who received at least 1 dose of study drug (IDELA or combination drugs). Per prespecified analysis, participants were grouped by disease (CLL, iNHL, MCL) and by treatment regimen (cohort).
Arm/Group | Idelalisib + Rituximab | Idelalisib + Bendamustine | Idelalisib + Everolimus | Idelalisib + Bortezomib | Idelalisib + Rituximab + Bendamustine | Idelalisib + Ofatumumab | Idelalisib + Fludarabine | Idelalisib + Chlorambucil | Idelalisib + Rituximab + Chlorambucil | Idelalisib + Rituximab + Lenalidomide
All-Cause Mortality (participants affected / at risk) | 1/51 | 6/51 | 4/18 | 3/18 | 1/33 | 4/21 | 2/12 | 0/15 | 3/15 | 2/7
Serious Adverse Events (participants affected / at risk) | 20/51 | 37/51 | 14/18 | 6/18 | 17/33 | 12/21 | 9/12 | 9/15 | 8/15 | 5/7
Other Adverse Events (participants affected / at risk) | 51/51 | 51/51 | 18/18 | 15/18 | 33/33 | 21/21 | 12/12 | 15/15 | 15/15 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib + Rituximab (N=51) | Idelalisib + Bendamustine (N=51) | Idelalisib + Everolimus (N=18) | Idelalisib + Bortezomib (N=18) | Idelalisib + Rituximab + Bendamustine (N=33) | Idelalisib + Ofatumumab (N=21) | Idelalisib + Fludarabine (N=12) | Idelalisib + Chlorambucil (N=15) | Idelalisib + Rituximab + Chlorambucil (N=15) | Idelalisib + Rituximab + Lenalidomide (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coombs positive haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 5 | 2 | 0 | 1 | 1 | 1 | 4 | 2 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endocrine disorder (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis microscopic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 2 | 1 | 0 | 1 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Generalised oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 10 | 1 | 1 | 5 | 2 | 1 | 1 | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspergillus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cytomegalovirus gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus viraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster disseminated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Human herpesvirus 6 infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Listeria sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Listeriosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mycobacterium avium complex infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Pneumonia (Infections and infestations) | 4 | 10 | 2 | 0 | 1 | 3 | 1 | 1 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia haemophilus (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib + Rituximab (N=51) | Idelalisib + Bendamustine (N=51) | Idelalisib + Everolimus (N=18) | Idelalisib + Bortezomib (N=18) | Idelalisib + Rituximab + Bendamustine (N=33) | Idelalisib + Ofatumumab (N=21) | Idelalisib + Fludarabine (N=12) | Idelalisib + Chlorambucil (N=15) | Idelalisib + Rituximab + Chlorambucil (N=15) | Idelalisib + Rituximab + Lenalidomide (N=7)
Anaemia (Blood and lymphatic system disorders) | 6 | 13 | 5 | 5 | 4 | 3 | 3 | 3 | 4 | 0
Coombs positive haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoglobulinaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 6 | 2 | 2 | 4 | 0 | 0 | 4 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 15 | 27 | 7 | 4 | 13 | 6 | 6 | 9 | 7 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 14 | 11 | 4 | 3 | 3 | 1 | 5 | 3 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 2 | 1 | 3 | 1 | 0 | 0 | 0 | 2
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Eyelid thickening (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 2 | 2 | 1 | 1 | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 10 | 6 | 1 | 3 | 3 | 2 | 1 | 1 | 3 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 11 | 2 | 3 | 8 | 4 | 2 | 2 | 6 | 6
Diarrhoea (Gastrointestinal disorders) | 20 | 14 | 9 | 7 | 12 | 11 | 6 | 6 | 8 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 9 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 3 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 5 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip blister (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 17 | 19 | 2 | 3 | 14 | 6 | 4 | 4 | 6 | 4
Noninfective gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 4 | 4 | 2 | 1 | 2 | 1 | 0 | 2 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 6 | 2 | 1 | 6 | 3 | 3 | 4 | 1 | 2
Asthenia (General disorders) | 5 | 4 | 3 | 2 | 2 | 1 | 2 | 0 | 2 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Chest pain (General disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0
Chills (General disorders) | 8 | 11 | 4 | 2 | 4 | 3 | 0 | 6 | 1 | 1
Face oedema (General disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 18 | 24 | 5 | 4 | 12 | 4 | 5 | 4 | 5 | 4
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Infusion site pain (General disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Injection site discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 2 | 3 | 3 | 0 | 2 | 1 | 2 | 0 | 1 | 1
Oedema (General disorders) | 1 | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 4 | 4 | 3 | 3 | 4 | 3 | 2 | 3 | 2 | 1
Pain (General disorders) | 5 | 4 | 3 | 2 | 3 | 0 | 2 | 3 | 2 | 0
Peripheral swelling (General disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 18 | 26 | 4 | 3 | 18 | 6 | 4 | 3 | 8 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Hypogammaglobulinaemia (Immune system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Seasonal allergy (Immune system disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Aspergillus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 0
Herpes virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 3 | 3 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0
Human herpesvirus 6 infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infected cyst (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mycobacterium avium complex infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 5 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 3 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Parvovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2 | 0 | 2 | 5 | 1 | 0 | 2 | 3 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 4 | 6 | 0 | 1 | 4 | 4 | 0 | 2 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 10 | 10 | 1 | 2 | 3 | 4 | 1 | 1 | 3 | 0
Urinary tract infection (Infections and infestations) | 3 | 3 | 2 | 1 | 2 | 3 | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 0 | 5 | 3 | 0 | 0 | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Traumatic ulcer (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 8 | 17 | 2 | 5 | 5 | 2 | 3 | 1 | 4 | 5
Aspartate aminotransferase increased (Investigations) | 8 | 14 | 2 | 5 | 3 | 2 | 3 | 1 | 3 | 5
Blood albumin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 6 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2
Blood creatinine increased (Investigations) | 1 | 1 | 4 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood immunoglobulin A decreased (Investigations) | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood immunoglobulin G decreased (Investigations) | 1 | 3 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Blood immunoglobulin M decreased (Investigations) | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 4 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 5
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Carbon dioxide decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 4 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Glucose tolerance increased (Investigations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 3 | 2 | 0 | 0 | 2 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Protein total decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 3 | 6 | 1 | 2 | 3 | 1 | 2 | 1 | 2 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 7 | 6 | 3 | 2 | 5 | 5 | 2 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 3 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 0 | 1 | 2 | 2 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 2 | 0 | 3 | 2 | 0 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 5 | 6 | 4 | 4 | 2 | 1 | 2 | 5 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0 | 2 | 0 | 2 | 0 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 6 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 4 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 5 | 3 | 0 | 1 | 3 | 1 | 1 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 | 0 | 1 | 4 | 1 | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 8 | 4 | 1 | 4 | 3 | 4 | 2 | 2 | 2 | 2
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 4 | 7 | 2 | 2 | 1 | 2 | 2 | 1 | 3 | 0
Headache (Nervous system disorders) | 12 | 4 | 3 | 0 | 3 | 2 | 2 | 2 | 1 | 2
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 0 | 3 | 0 | 2 | 1 | 3 | 3 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 7 | 11 | 3 | 0 | 6 | 2 | 1 | 4 | 3 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 3 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Genital swelling (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 18 | 7 | 0 | 9 | 9 | 6 | 7 | 4 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 9 | 3 | 0 | 5 | 7 | 2 | 3 | 3 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 7 | 0 | 0 | 1 | 2 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 1 | 0 | 1 | 0 | 2 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 2 | 0 | 2 | 1 | 0 | 0 | 1 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 2 | 1 | 1 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 3 | 0 | 3 | 3 | 1 | 0 | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 3 | 0 | 0 | 1 | 3 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 2 | 2 | 0 | 1 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Actinic elastosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 0
Lentigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 6 | 7 | 2 | 2 | 1 | 0 | 1 | 3 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 6 | 4 | 2 | 5 | 1 | 0 | 1 | 2 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 11 | 16 | 5 | 5 | 13 | 4 | 2 | 3 | 5 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 2 | 4 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 2 | 3 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 2 | 0 | 1 | 3 | 2 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 2 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years